CLINICAL TRIAL: NCT05867823
Title: Effectivity of an Occupational-self-analysis Intervention Through a Mobile Application (OcupApp) in People With Anxiety or Depression: A Randomised Controlled Trial Protocol
Brief Title: OcupApp: Occupational Self-analysis Intervention Through an Mobile Application
Acronym: OcupApp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Collaborators: University of Vic - Central University of Catalonia (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, María Rodríguez Bailón, "OcupApp": Development and effectiveness of a mobile application for the involvement in meaningful activities in the elderly population., University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1-2020_25
Record Dates: First submitted 2023-05-08; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Anxiety Disorder; Depressive Disorder; Occupational Therapy; Mobile App
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking will be single blind since the researchers will know the assigned arm. Participants will know the group they belong, but not the hypotheses of the study or the superiority that is sought of one intervention over the other. However, data evaluators will remain blind to the allocation of patients to group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OcuApp Users (Experimental): the experimental group will use a movile aplication (OcuApp), to generate a personal self-analisys about meaningful activities.
  Interventions: Behavioral: OcuApp
- Three-part work users (Active Comparator): The intervention on the control group will focus on offering to the participants an informative three-part work on the positive effects of performing activities.
  Interventions: Behavioral: Three-part work

INTERVENTIONS:
Behavioral: OcuApp — The participants will have instaled a mobile aplication (OcuApp) by a member of the researchs team who will teach them how to use it. The person must register the activities they carry out throughout a week and mark each one of them with a punctuation (from 1 to 5) related to the meaning of the following dimensions: identity, pleasure, competence, importance and value of the activity by other people.The application also allows to collect other information such as where the activity takes place, its duration, and the people with whom it is carried out. Also, at the end of the week, the application will ask users about their perceived occupational balance. All the information registered in the mobile application will be returned to the person in a dynamic and understandable way. Based on this, the person can establish two goals to accomplish. In this sense, OcupApp will offer personalized recommendations based on the objectives to be achieved related to the dimensions of meaning.
  Arms: OcuApp Users
Behavioral: Three-part work — The intervention on the control group will focus on offering to the participants an informative three-part work on the positive effects of performing activities to control anxiety and depression. After providing this information, any doubts in this regard will be answered.
  Arms: Three-part work users

SUMMARY:
The goal of this clinical trial is to test the effectiveness of the use of mobile application ("OcupApp") to generate a personal self-analysis about meaningful activities in which adults between the ages of 50 and 70 with anxiety and subclinical depression participant.

A randomized study will be carried out comparing the effects of the use of the application "OcupApp" with a control intervention on the quality of life related to health, mental health, frequency of participation on meaningful activities, and perceived occupational balance.

DETAILED DESCRIPTION:
OcupApp is a mobile application developed within the research team, which aims to promote occupational self-analysis in adults with depression and/or anxiety. The mobile application allows to offer feedback to participants about the meaning of the activities they carry out daily and their perception of occupational balance, which generates a subjective self-reflection that can lead to the implementation of some personal changes in their weekly routine. For this, the person must register the activities they carry out throughout a week and mark each one of them with a punctuation related to the meaning of the following dimensions: identity, pleasure, competence, importance and value of the activity by other people. The punctuation give will be on a Likert-type scale from 1 to 5. The application also allows to collect other information such as where the activity takes place, its duration, and the people with whom it is carried out. Also, at the end of the week, the application will ask users about their perceived occupational balance. All the information registered in the mobile application will be returned to the person in a dynamic and understandable way. Based on this, the person can establish two goals to accomplish. In this sense, OcupApp will offer personalized recommendations based on the objectives to be achieved related to the dimensions of meaning.

ELIGIBILITY:
Inclusion Criteria:

* Have a smarthphone and know how to use mobile apps to exchange information.
* Have a low or moderate depression (DEP 5 <= 4) or low or moderate anxiety (ANX5 <= 3) or DEP5 or ANX5 =3).

Exclusion Criteria:

* Have a serious mental illness or psychosis.
* Have a diagnosis of dementia
* Have language problems or cognitive alterations that doesn't allow comprehension of assessment tools.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The World Health Organization Quality of Life (WHOQOL-BREF) | 15 minutes
  The WHOQOL is a generic, multidimensional profile for assessing quality of life with 26 questions; 2 related to their general quality of life and their satisfaction with their health status and 24 item-version assessing 4 domains of quality of life (physical health, psychological health, social relations and environment).

SECONDARY OUTCOMES:
The General Health Questionnaire (GHQ). | 10 minutes
  The mental health of the participants was assessed using the 12-item version of the General Health Questionnaire (GHQ), which is a valid and reliable instrument to assess psychological well-being and distinct aspects of distress.The total sum of scores can range from 0 to 36, with higher total scores reflecting higher levels of psychological distress.

OTHER OUTCOMES:
The Engagement in Meaningful Activities Survey (EMAS). | 5 minutes
  The 12 items comprising the EMAS measure engagement in meaningful activities by assessing through a 5-point Likert-scale varied aspects of meaning such as creativity, pleasure, and satisfaction, feelings of competence and control, and a sense of belonging and a capacity for helping others.
Occupational Balance Questionnaire (OBQ). | 15 minutes
  The Occupational Balance Questionnaire (OBQ) is a questionnaire in which the person evaluates their occupational balance in relation to their current situation and their daily life. a final score can be obtained summing scores from 0 to 65, where a higher score indicates a higher Occupational balance.

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published in an indexed journal. Once collected, participants' data will be uploaded to a public repository.
Supporting Information: Study Protocol
Time Frame: The protocol will be accessible when published in a journal and the data once collected.
Access Criteria: Public